CLINICAL TRIAL: NCT04102111
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Platform Study Evaluating the Efficacy and Safety of Interventions in Participants With Moderately to Severely Active Crohn's Disease
Brief Title: A Study Evaluating Participants With Moderately to Severely Active Crohn's Disease
Acronym: PRISM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IAC completed review of futility analysis data & determined that futility criteria were met. As a result, Janssen made decision to stop trial immediately.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR108455; 2018-000649-38 (EudraCT Number); 67864238PACRD2001 (Other: Janssen Research & Development, LLC); PLATFORMPACRD2001 (Other: Janssen Research & Development, LLC); 2019-003335-37 (EudraCT Number)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Results first posted 2022-12-09 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- JNJ-67864238 (Experimental): Participants will receive oral tablets of JNJ-67864238 twice daily for 12 weeks.
  Interventions: Drug: JNJ-67864238
- Placebo (Placebo Comparator): Participants will receive oral tablets of matching placebo twice daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-67864238 — Participants will receive oral tablets of JNJ-67864238 twice daily.
  Arms: JNJ-67864238
Drug: Placebo — Participants will receive oral tablets of matching placebo twice daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of JNJ-active as measured by the change in the Crohn's Disease Activity Index (CDAI) score and Simplified Endoscopic Score for Crohn's disease (SES-CD) from baseline at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Have active Crohn's disease, defined as a baseline Crohn's Disease Activity Index (CDAI) score of greater than or equal to (>=) 220 and less than or equal to (<=) 450
* Have evidence of active ileocolonic Crohn's disease as assessed by an Simplified Endoscopic Score for Crohn's disease (SES-CD) score >=3 at screening by central endoscopy reading; or an elevated screening C-reactive protein (CRP) (greater than [>] 0.3 milligrams per deciliter [mg/dL] or 3.0 milligrams per liter [mg/L]) or an elevated screening fecal calprotectin (>250 micrograms per mg [mcg/mg])
* A participant with a family history of colorectal cancer, personal history of increased risk of colorectal cancer, age > 50 years, or other known risk factor must be up-to-date on colorectal cancer surveillance (may be performed during screening). Adenomatous polyps must be removed before the first administration of the study intervention
* A woman of childbearing potential must have a negative highly sensitive serum (Beta-human chorionic gonadotropin [beta-hCG]) pregnancy test result at screening and a negative urine pregnancy test result at Week 0
* Has previously demonstrated inadequate response to, loss of response to, or intolerance to an approved biologic therapy (unless otherwise specified in the JNJ-67864238 intervention cohort specific criteria, that is, anti-tumor necrosis factor (TNF) alpha agents (for example, infliximab, adalimumab, certolizumab pegol], anti- interleukin (IL)-12/23 agents [for example, ustekinumab], or anti-integrin agents [for example, vedolizumab]) or has previously demonstrated an inadequate response to or failed to tolerate corticosteroids or immunomodulators (that is, 6-mercaptopurine [6-MP], azathioprine [AZA], and methotrexate [MTX]) but not a biologic, that is, the biologic nonfailures (Bio-NF) population
* Therapy for the treatment of Crohn's disease must include at least 1 of the following medications, which should have been maintained at stable doses prior to the baseline (Week 0) visit: (a) Oral 5-aminosalicylic acid (5-ASA) compounds; (b) Oral corticosteroids at a prednisone-equivalent dose <= 25 milligrams per day (mg/day), or 9 mg/day of budesonide, or 5 mg/day beclomethasone dipropionate; (c) Antibiotics being used as a primary treatment of Crohn's disease; and (d) Conventional immunomodulators (that is, AZA, 6-MP, or MTX) if participants have been taking them for at least 12 weeks and have been at a stable dose for at least 4 weeks prior to baseline

Exclusion Criteria:

* Prior exposure to an anti-IL-12/23 (that is ustekinumab) or anti-IL-23 agents or related compound (including risankizumab, brazikumab, guselkumab, mirikizumab, and related compounds). Exception is made for participants who have had minimal exposure to ustekinumab at its approved labeled dosage and have met the required wash-out criteria and have not demonstrated inadequate response or intolerance to ustekinumab
* Known allergies, hypersensitivity, or intolerance to JNJ-67864238 or its excipients
* Has complications of Crohn's disease such as symptomatic strictures or stenoses, short gut syndrome, or any other manifestation that might be anticipated to require surgery, could preclude the use of the CDAI to assess response to therapy, or would possibly confound the ability to assess the effect of treatment with JNJ-67864238
* Has had any kind of bowel resection within 6 months or any other intra-abdominal surgery within 3 months before baseline
* Initiation of total (complete) or partial (supplemental) parenteral nutrition administered through any indwelling catheter less than (<) 3 weeks before baseline or anticipated to require parenteral nutrition administered through an indwelling catheter during enrollment in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (63):
- United States (13):
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Gastro Florida, Clearwater, Florida
  - Gastroenterology Associates of Central GA, Macon, Georgia
  - CroNOLA, LLC, Houma, Louisiana
  - Washington University, St Louis, Missouri
  - NYU Langone Long Island Clinical Research Associates, Lake Success, New York
  - Columbia University Medical Center, New York, New York
  - Northshore Gastroenterology Research, LLC, Beachwood, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Northshore Gastroenterology Research, LLC, Westlake, Ohio
  - Digestive Disease Specialists Inc, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Gastroenterology Research of San Antonio, San Antonio, Texas
- Argentina (6):
  - Cer Instituto Medico, Buenos Aires
  - CINME Centro de Investigaciones Metabolicas, CABA
  - Clinica Adventista Belgrano, Ciudad de Buenos Aires
  - Sanatorio Duarte Quiroz, Córdoba
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Fundacion de Estudios Clinicos, Rosario
- Germany (4):
  - Universitatsklinikum Schleswig Holstein Kiel, Kiel
  - Eugastro GmbH, Leipzig
  - Universitaetsklinikum Mannheim, Mannheim
  - Universitaetsklinikum Ulm, Klinik fuer Innere Medizin II, Ulm
- Italy (14):
  - Policlinico di Bari Ospedale Giovanni XXIII, Bari
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Ospedaliera G. Brotzu, Cagliari
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Ospedale Classificato Equiparato Sacro Cuore Don Calabria di Negrar, Negrar ( Ve)
  - Ospedale Maggiore della Carita, Novara
  - Azienda Ospedaliera di Padova, Padua
  - IRCCS Policlinico San Matteo, Università degli studi di Pavi, Pavia
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Azienda Ospedaliera G.Salvini Ospedale di Rho, Rho
  - Policinico A Gemelli, Roma
  - Istituto Clinico Humanitas, Rozzano
  - A.O.Citta della Salute e della Scienza di Torino, Torino
- Poland (5):
  - Gastromed Kralisz Romatowski Stachurska Sp. j., Bialystok
  - Endoskopia Sp z o.o., Sopot
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centralny Szpital Kliniczny Mswia, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
- Russia (11):
  - Immanuel Kant Baltic Federal University, Kaliningrad
  - Kemerovo Region Clinical Hospital, Kemerovo
  - City Hospital #13 of Avtozavodsky, Nizhny Novgorod
  - Medical Center SibNovoMed LLC, Novosibirsk
  - Rostov State Medical University (RSMU) based on City Hospital No. 20, Rostov-on-Don
  - International Medical Centre SOGAZ, Saint Petersburg
  - City Hospital named after St. Martyr Elizabeth, Saint Petersburg
  - Non State Healthcare Inst. Railway Clinical Hospital at Samara station JSC 'Russian Railways', Samara
  - GBUZ Respublican Clinical Hospital n.a. GG Kuvatova, Ufa
  - Medical diagnostic centre LTD 'MDC', Yaroslavl
  - Medical Center Meditsinskie Tekhnologii, Yekaterinburg
- Ukraine (10):
  - MNCE City Clinical Hospital No 2 named after prof O O Shalimov of the Kharkiv City Council, Kharkiv
  - GI L.T.Malaya Therapy National Institute of the NAMS of Ukraine, Kharkiv
  - Kyivska miska klinichna likarnia 18, Kyiv
  - Medical Center 'Ok Clinic' of International Institute of Clinical Research LLC, Kyiv
  - Danylo Halytsky Lviv National Medical University, Lviv
  - Municipal Non-profit Enterprise 'Odesa Regional Clinical Hospital' Odesa Regional Council, Odesa
  - Municipal Non-commercial Enterprise Ternopil University Hospital of Ternopil Regional Council, Ternopil
  - MNCE Zakarpatska Regional Clinical Hospital named after A Novak of Zakarpatska Regional Council, Uzhhorod
  - Medical Center Ltd 'Health Clinic', Vinnytsia
  - VNMUn.af.Pyrogova,CNE Vinnytsia Regional Clinical Hospital n.af.Pyrogova Vinnytsia Regional Council, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants were randomized to receive matching placebo tablets orally twice daily for 12 weeks.
- JNJ-67864238: Participants were randomized to receive JNJ-67864238 300 milligrams (mg) tablets orally twice daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | JNJ-67864238
Started | 18 | 30
Completed | 14 | 23
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Study terminated by sponsor | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | JNJ-67864238 | Total
Number analyzed (Participants) | 18 | 30 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (8.72) | 37.7 (13.49) | 38.4 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 21
  Male | 11 | 16 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 18 | 29 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 0 | 1 | 1
  ITALY | 2 | 4 | 6
  POLAND | 2 | 3 | 5
  RUSSIAN FEDERATION | 8 | 10 | 18
  UKRAINE | 4 | 10 | 14
  UNITED STATES | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Crohn's Disease Activity Index (CDAI) Score at Week 12
Description: CDAI is a validated measure of illness severity derived as sum of 8 different Crohn's disease (CD)-related variables (extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s)/opiates, and general well-being). Last 3 variables were scored over 7 days by participant on diary card. Score ranges from 0 to 600; higher score=higher disease activities. Participants who had incomplete data (less than or equal to [<=]4 component values missing) at the visit, had their last available component value carried forward to calculate CDAI Score. Participants who had prohibited change in concomitant CD medication, CD-related surgery or discontinued intervention due to lack of efficacy or adverse event of worsening CD prior to Week 12 had their baseline value carried forward. Participants who had discontinuation of intervention due to corona virus disease-19 related reasons had their CDAI data as missing.
Time Frame: Baseline and Week 12
Population: Full analysis set (FAS) included participants who were randomized to either JNJ-67864238 or placebo and received at least 1 dose of study intervention. Here, 'N' (Number of participants analyzed) included all participants evaluable for this outcome measure (OM).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | JNJ-67864238
Number analyzed (Participants) | 15 | 23
units on a scale | -153.2 (94.71) | -124.6 (124.94)
Statistical Analysis 1: Comparison: Placebo vs JNJ-67864238; Test type: Other; p = 0.288, Mixed Model for Repeated Measures (MMRM); Least Squares Means = 37.4, 90% CI 2-sided [-21.0 to 95.8]

2. Secondary Outcome: Change From Baseline in Simplified Endoscopic Score for Crohn's Disease (SES-CD) at Week 12
Description: SES-CD scoring system assesses disease severity in participants with CD. It is based on evaluation of 4 endoscopic components (presence/size of ulcers, proportion of mucosal surface covered by ulcers, proportion of mucosal surface affected by any lesions and presence/type of narrowing [strictures/ stenosis clinically] across 5 predefined ileocolonic segments (ileum, right colon, transverse colon, left colon and rectum). Each component score= 0 to 3 for each segment, total score calculated as sum of all component scores for all segments. Maximum sub-score for narrowings=11 points. Total SES-CD score ranges=0 to 56, where higher scores=more severe disease. Participants who had prohibited change in concomitant CD medication, CD-related surgery or discontinued intervention due to lack of efficacy/AE of worsening CD prior to Week 12 had their baseline value carried forward. Participants who had discontinuation of intervention due to COVID-19 related reasons had their CDAI data as missing.
Time Frame: Baseline and Week 12
Population: FAS included participants who were randomized to either JNJ-67864238 or placebo and received at least 1 dose of study intervention. Here, 'N' (Number of participants analyzed) included all participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | JNJ-67864238
Number analyzed (Participants) | 14 | 22
units on a scale | -0.4 (2.27) | -1.6 (4.50)

3. Secondary Outcome: Percentage of Participants With Clinical Response at Week 12
Description: Percentage of participants with clinical response at Week 12 were reported. Clinical response is defined as a greater than or equal to (>=) 100-point reduction from baseline in CDAI score or CDAI score less than (<) 150. The CDAI is a validated multi-item measure of severity of illness derived as a weighted sum of 8 different Crohn's disease-related variables (extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being). The last 3 variables were scored over 7 days by the participant on a diary card. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities.
Time Frame: Week 12
Population: FAS included participants who were randomized to either JNJ-67864238 or placebo and received at least 1 dose of study intervention. Participants who met 1 or more treatment failure rules: had prohibited change in concomitant CD medication, had CD-related surgery, discontinued intervention due to lack of efficacy or AE of worsening CD prior to Week 12 or discontinuation of intervention due to COVID-19 related reasons, were not considered to be in clinical response.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-67864238
Number analyzed (Participants) | 18 | 30
percentage of participants | 61.1 | 46.7

4. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 12
Description: Percentage of participants with clinical remission at Week 12 were reported. Clinical remission is defined as CDAI score <150. The CDAI is a validated multi-item measure of severity of illness derived as a weighted sum of 8 different Crohn's disease-related variables (extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stools, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being). The last 3 variables were scored over 7 days by the participant on a diary card. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities.
Time Frame: Week 12
Population: FAS included participants who were randomized to either JNJ-67864238 or placebo and received at least 1 dose of study intervention. Participants who met 1 or more treatment failure rules: had prohibited change in concomitant CD medication, had CD-related surgery, discontinued intervention due to lack of efficacy or AE of worsening CD prior to Week 12 or discontinuation of intervention due to COVID-19 related reasons, were not considered to be in clinical remission.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-67864238
Number analyzed (Participants) | 18 | 30
percentage of participants | 44.4 | 40.0

5. Secondary Outcome: Percentage of Participants With Patient-reported Outcome (PRO)-2 Remission at Week 12
Description: Percentage of participants with PRO-2 remission at Week 12 were reported. PRO-2 remission is defined as abdominal pain (AP) mean daily score (AP component of the CDAI) <=1 and stool frequency (SF) mean daily score of <=3, that is, AP <=1 and SF <=3. PRO-2 is a composite index consisting of weighted scoring of both variables. PRO-2 scores range from 0 to no upper limit with higher scores indicating more severe disease.
Time Frame: Week 12
Population: FAS included participants who were randomized to either JNJ-67864238 or placebo and received at least 1 dose of study intervention. Participants who met 1 or more treatment failure rules: had prohibited change in concomitant CD medication, had CD-related surgery, discontinued intervention due to lack of efficacy or AE of worsening CD prior to Week 12 or discontinuation of intervention due to COVID-19 related reasons, are not considered to be PRO-2 remission.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-67864238
Number analyzed (Participants) | 18 | 30
percentage of participants | 33.3 | 33.3

6. Secondary Outcome: Percentage of Participants With Endoscopic Response at Week 12
Description: Endoscopic response is defined as at least 50 percent (%) improvement from baseline in SES-CD score. SES-CD scoring system assesses disease severity in participants with CD. It is based on evaluation of 4 endoscopic components (presence/size of ulcers, proportion of mucosal surface covered by ulcers, proportion of mucosal surface affected by any lesions and presence/type of narrowing [strictures/ stenosis clinically] across 5 predefined ileocolonic segments (ileum, right colon, transverse colon, left colon and rectum). Each component score=0 to 3 for each segment, total score calculated as sum of all component scores for all segments. Maximum sub-score for narrowings=11 points. Total SES-CD score range=0 to 56, where higher score=more severe disease.
Time Frame: Week 12
Population: FAS included participants who were randomized to either JNJ-67864238 or placebo and received at least 1 dose of study intervention. Participants who met 1 or more treatment failure rules: had prohibited change in concomitant CD medication, had CD-related surgery, discontinued intervention due to lack of efficacy or AE of worsening CD prior to Week 12 or discontinuation of intervention due to COVID-19 related reasons, are not considered to be in endoscopic response.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-67864238
Number analyzed (Participants) | 18 | 30
percentage of participants | 5.6 | 26.7

7. Secondary Outcome: Percentage of Participants With Endoscopic Remission at Week 12
Description: Endoscopic remission defined as an SES-CD score of <=2. SES-CD scoring system assesses disease severity in participants with CD. It is based on evaluation of 4 endoscopic components (presence/size of ulcers, proportion of mucosal surface covered by ulcers, proportion of mucosal surface affected by any lesions and presence/type of narrowing [strictures/ stenosis clinically] across 5 predefined ileocolonic segments (ileum, right colon, transverse colon, left colon and rectum). Each component score=0 to 3 for each segment, total score calculated as sum of all component scores for all segments. Maximum sub-score for narrowings=11 points. Total SES-CD score range=0 to 56, where higher score=more severe disease.
Time Frame: Week 12
Population: FAS included participants who were randomized to either JNJ-67864238 or placebo and received at least 1 dose of study intervention. Participants who met 1 or more treatment failure rules: had prohibited change in concomitant CD medication, had CD-related surgery, discontinued intervention due to lack of efficacy or AE of worsening CD prior to Week 12 or discontinuation of intervention due to COVID-19 related reasons, are not considered to be in endoscopic remission.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | JNJ-67864238
Number analyzed (Participants) | 18 | 30
percentage of participants | 5.6 | 16.7

ADVERSE EVENTS:
Time Frame: Up to 12 weeks for serious and other (non-serious) adverse events and up to 16 weeks for all-cause mortality
Description: The safety analysis set included all randomized participants who received at least 1 dose of study intervention (placebo or JNJ-67864238).
Arm/Group | Placebo | JNJ-67864238
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/18 | 4/30
Other Adverse Events (participants affected / at risk) | 9/18 | 14/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | JNJ-67864238 (N=30)
Crohn's Disease (Gastrointestinal disorders) | 1 | 2
Covid-19 (Infections and infestations) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | JNJ-67864238 (N=30)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Basophilia (Blood and lymphatic system disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Crohn's Disease (Gastrointestinal disorders) | 2 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 1
Gastritis Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Mouth Swelling (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Oral Disorder (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Hepatic Cyst (Hepatobiliary disorders) | 1 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 1 | 0
Clostridium Difficile Infection (Infections and infestations) | 0 | 1
Covid-19 (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Pyoderma (Infections and infestations) | 0 | 1
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Lymphocyte Count Decreased (Investigations) | 2 | 0
Neutrophil Count Decreased (Investigations) | 0 | 1
Hypoferritinaemia (Metabolism and nutrition disorders) | 1 | 0
Haemangioma of Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness Exertional (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 4
Sciatica (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal Swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT04102111/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/11/NCT04102111/SAP_001.pdf